CLINICAL TRIAL: NCT02208271
Title: A Validated Necrosis Assay to Determine the Need for Revision Surgery in Metal-on-metal Total Hip Arthroplasty
Status: Suspended | Type: Observational
Why Stopped: The lab was acquired by another company and has put this study's samples on hold.
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Collaborators: Charlotte Orthopedic Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HK003-14014
Record Dates: First submitted 2014-07-17; First posted 2014-08-05 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Arthritis, Failure of Total Hip
Keywords: tissue necrosis; metal on metal total hip; biomarker
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control: pre-operative total hip patients with no existing total hip implant
- Metal on polyethylene: patients who have a failed metal on polyethylene total hip implant and are presenting for revision surgery
- Metal on Metal: patients who have a failed metal on metal total hip implant and are presenting for revision surgery

SUMMARY:
The purpose of the study is to develop a biomarker assay to be used as a diagnostic tool for adverse local tissue reaction, or tissue necrosis, in a metal on metal total hip replacement.

A convenience sample of a total of 100 hip patients will be enrolled: 50 metal-on-metal revision hips, 25 metal-on-poly revision hips, and 25 pre-operative total hips (no implant, control group) will be enrolled. Preoperative blood serum samples and intraoperative synovial fluid will be obtained from all hips and used for biomarker testing. Additionally, intraoperative assessment of tissue necrosis will be assessed.

DETAILED DESCRIPTION:
Well-functioning MoM implants have shown an increase in serum cobalt and chromium (CoCr) ion levels from the metal debris generated from the implant wear.However, the current evidence suggests that measuring ion levels is unreliable and that increasing ion levels do not correlate with tissue damage. In addition to measuring blood and synovial fluid metal ion levels, ultrasound and MRI with metal artifact reduction sequences (MARS) have been utilized to assess periarticular reactions secondary to metal wear debris. Despite metal reduction software these scans are frequently difficult to interpret. While each of these tests has merit, at the present time there is no single diagnostic test available which delineates the key issue that demands urgent surgical intervention, i.e. tissue necrosis. It is important to have a reliable test to guide surgeons and patients in the shared decision-making process of when surgical intervention is necessary to prevent disabling tissue damage. For this reason, the current study proposes an examination of preoperative serum samples of subjects in addition to synovial fluid collected during revision surgery for biomarkers that may indicate tissue necrosis. To maximize the chance of success of identifying serum biomarkers, all samples will be analyzed using multianalyte assay, biomarker tests. The purpose of the study is to develop a biomarker assay to be used as a diagnostic tool for adverse local tissue reaction, or tissue necrosis, in a metal on metal total hip replacement.

A convenience sample of a total of 100 hip patients will be enrolled: 50 metal-on-metal revision hips, 25 metal-on-poly revision hips, and 25 pre-operative total hips (no implant, control group) will be enrolled. Preoperative blood serum samples and intraoperative synovial fluid will be obtained from all hips and used for biomarker testing. Additionally, intraoperative assessment of tissue necrosis will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for a metal on metal hip revision who have cobalt and chromium metal ion levels tested within 6 months of the date of the planned revision surgery.
* Patients presenting for a metal on poly hip revision
* Revision hip patients must be greater than one year postoperative
* The diagnosis at the time of the index, or primary, hip replacement was osteoarthritis.
* Patients who have hip osteoarthritis but have not had a total hip surgery (control)

Exclusion Criteria:

* Patients presenting for a metal on metal hip revision who have cobalt and chromium metal ion levels tested >6 months of the date of the planned revision
* Patients with a total hip on the contralateral side.
* Patients with a prior history of periprosthetic infection
* Revision cases where the diagnosis at the time of the index, or primary, hip replacement was not osteoarthritis.
* Prisoners
* Patients not willing to consent for the proposed treatment
* Patients with an altered mental status
* Active, concurrent metastatic infection
* Active, superficial infection
* Patients presenting for a metal on poly hip revision to treat trunionosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A convenience sample of a total of 100 hip patients will be enrolled at orthopedic clinics.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of patients with serum and synovial fluid biomarkers | participants will be followed for the duration of their hospital stay, an expected average of 2 hours
  Blood Serum and Synovial fluid will be tested using a multi-analyte assay test

SECONDARY OUTCOMES:
The number of patients with tissue necrosis | participants will be followed for the duration of their hospital stay, an expected average of 2 hours
  Tissue necrosis will be assessed during total hip surgery.
  Tissue necrosis will be scored in subsets including: intraoperative tissue damage, histological necrosis score, histologic ALVAL score, inflammatory infiltrate, and tissue organization

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Fehring, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina, Charlotte, North Carolina, United States

REFERENCES:
- [Background] MacDonald SJ. Metal-on-metal total hip arthroplasty: the concerns. Clin Orthop Relat Res. 2004 Dec;(429):86-93. doi: 10.1097/01.blo.0000150309.48474.8b. PMID 15577471
- [Background] Lindgren JU, Brismar BH, Wikstrom AC. Adverse reaction to metal release from a modular metal-on-polyethylene hip prosthesis. J Bone Joint Surg Br. 2011 Oct;93(10):1427-30. doi: 10.1302/0301-620X.93B10.27645. PMID 21969447
- [Background] Lombardi AV Jr, Barrack RL, Berend KR, Cuckler JM, Jacobs JJ, Mont MA, Schmalzried TP. The Hip Society: algorithmic approach to diagnosis and management of metal-on-metal arthroplasty. J Bone Joint Surg Br. 2012 Nov;94(11 Suppl A):14-8. doi: 10.1302/0301-620X.94B11.30680. PMID 23118373
- [Background] Cobb AG, Schmalzreid TP. The clinical significance of metal ion release from cobalt-chromium metal-on-metal hip joint arthroplasty. Proc Inst Mech Eng H. 2006 Feb;220(2):385-98. doi: 10.1243/09544119JEIM78. PMID 16669404
- [Background] Mabilleau G, Kwon YM, Pandit H, Murray DW, Sabokbar A. Metal-on-metal hip resurfacing arthroplasty: a review of periprosthetic biological reactions. Acta Orthop. 2008 Dec;79(6):734-47. doi: 10.1080/17453670810016795. PMID 19085489
- [Background] Tower SS. Arthroprosthetic cobaltism: neurological and cardiac manifestations in two patients with metal-on-metal arthroplasty: a case report. J Bone Joint Surg Am. 2010 Dec 1;92(17):2847-51. doi: 10.2106/JBJS.J.00125. Epub 2010 Oct 29. No abstract available. PMID 21037026
- [Background] Campbell P, Ebramzadeh E, Nelson S, Takamura K, De Smet K, Amstutz HC. Histological features of pseudotumor-like tissues from metal-on-metal hips. Clin Orthop Relat Res. 2010 Sep;468(9):2321-7. doi: 10.1007/s11999-010-1372-y. PMID 20458645
- [Background] Leopold SS, Berger RA, Patterson L, Skipor AK, Urban RM, Jacobs JJ. Serum titanium level for diagnosis of a failed, metal-backed patellar component. J Arthroplasty. 2000 Oct;15(7):938-43. doi: 10.1054/arth.2000.6632. PMID 11061457
- [Background] Griffin WL, Fehring TK, Kudrna JC, Schmidt RH, Christie MJ, Odum SM, Dennos AC. Are metal ion levels a useful trigger for surgical intervention? J Arthroplasty. 2012 Sep;27(8 Suppl):32-6. doi: 10.1016/j.arth.2012.03.020. Epub 2012 May 17. PMID 22608683